CLINICAL TRIAL: NCT00321932
Title: A Randomized Phase II of Zoledronic Acid (Zometa) in the Prevention of Osteoporosis in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Zoledronic Acid in Preventing Osteoporosis in Patients Undergoing Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005NT018; UMN-0506M70866 (Other: IRB, University of Minnesota); UMN-MT2005-06 (Other: Blood and Marrow Transplantation Program); NOVARTIS-CZOL446EUS29 (Other: Novartis)
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Osteoporosis; Ovarian Cancer
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Osteoporosis; Ovarian Neoplasms | interventions — Calcium; Calcium Carbonate; Calcium Citrate; Calcium Gluconate; Cholecalciferol; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (control) (Active Comparator): Patients receive oral cholecalciferol (vitamin D) and oral calcium once a day for 12 months.
  Interventions: Dietary Supplement: calcium; Dietary Supplement: cholecalciferol
- Arm II (treatment) (Experimental): Patients receive vitamin D and calcium as in arm I. Patients also receive zoledronic acid intravenously (IV) over 15-30 minutes at 28 days prior to stem cell transplantation and at 3 and 6 months after transplantation.
  Interventions: Dietary Supplement: calcium; Dietary Supplement: cholecalciferol; Drug: zoledronic acid

INTERVENTIONS:
Dietary Supplement: calcium — All randomized patients (control and study drug) will take 1000 mg of calcium and 400 - 500 International Units (IU) of vitamin D orally each day, beginning as soon as possible after study enrollment. These supplements may be taken either in the morning or in the evening with food. Participants will continue taking the supplements on a daily basis until the final study visit (approximately 12 months after the transplant date).
  Other Names: calcium carbonate; calcium citrate; calcium gluconate
Dietary Supplement: cholecalciferol — Given orally
Drug: zoledronic acid — Zoledronic acid (Zometa®) will be administered after randomization (but within 28 days prior to transplant) and at 3 and 6 months after the transplant for a total of 3 doses. The dose of Zometa will be 4 mg intravenous in 100 ml of sterile 0.9% sodium chloride, United States Pharmacopeia (USP), or 5% dextrose, USP infused over a minimum of 15 minutes for patients with a calculated creatinine clearance of ≥60 mL/min. The drug may be administered through a peripheral or a central intravenous line.
  Other Names: Zometa(R)
  Arms: Arm II (treatment)

SUMMARY:
RATIONALE: Zoledronic acid, vitamin D, and calcium may prevent bone loss in patients who are undergoing donor stem cell transplant.

PURPOSE: This randomized phase II trial is studying how well zoledronic acid works in preventing osteoporosis in patients undergoing donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate whether prophylactic administration of zoledronic acid can reduce the severity of bone mineral loss in patients undergoing allogeneic hematopoietic stem cell transplantation.

Secondary

* Determine the safety of zoledronic acid in these patients.

OUTLINE: This is a multicenter, open-label, prospective, randomized, controlled study. Patients are stratified according to participating center and type of transplant (myeloablative vs nonmyeloablative). Patients are randomized to 1 of 2 treatment arms.

* Arm I (control): Patients receive oral cholecalciferol (vitamin D) and oral calcium once a day for 12 months.
* Arm II (treatment): Patients receive vitamin D and calcium as in arm I. Patients also receive zoledronic acid intravenously (IV) over 15-30 minutes at 28 days prior to stem cell transplantation and at 3 and 6 months after transplantation.

In both arms, treatment continues in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥18 years
* Undergoing allogeneic hematopoietic stem cell transplantation (HCT) from any stem cell source with either a myeloablative or non-myeloablative conditioning regimen
* Bone mineral density measured by baseline pre-transplant DEXA scan in the osteopenic range (defined as a T-score between -1 and -2.5 standard deviation (SD) at either the lumbar spine or the proximal femur or both)
* Adequate renal function defined as: Calculated creatinine clearance of ≥ 60 ml/min using the Cockcroft-Gault formula:
* Serum calcium (corrected) of ≤ 10.5 mg/dl
* Patients (male or female) of reproductive potential are required to use a medically acceptable contraception while receiving zoledronic acid (if assigned study drug).
* Normal dental exam within the year prior to study registration
* Informed signed consent to participate in the study

Exclusion Criteria:

* Pre-existing metabolic bone disease including osteomalacia, hyperparathyroid bone disease, osteogenesis imperfecta, Paget's disease, rickets, or hypoparathyroidism.
* Multiple myeloma
* History of nontraumatic vertebral compression fractures
* History of the following endocrine disorders - hyperparathyroidism, hyperthyroidism.
* Malabsorption syndrome including Crohn's disease.
* Chronic liver disease
* Concomitant regular use of phenytoin.
* Known hypersensitivity to zoledronic acid (Zometa) or other biphosphonates
* Biphosphonate therapy within the preceding six months.
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants)
* Not pregnant or breastfeeding since zoledronic acid is classified as Pregnancy Category C: risk in pregnancy cannot be ruled out. A negative pregnancy test is required within 7 days of registration if pre- or perimenopausal (i.e., last menstrual period within one year of registration). Because it is not known whether zoledronic acid is excreted in breast milk, breastfeeding is not permitted while receiving study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-07; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda J. Burns, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing allogeneic hematopoietic stem cell transplantation (HCT) at participating institutions were offered this trial. If the patient met study requirements, the patient was registered and randomized.
Groups:
- Arm I (Standard of Care): Patients receive oral cholecalciferol (vitamin D) and oral calcium once a day for 12 months.
- Arm II (Treatment With Zometa): Patients receive vitamin D and calcium as in arm I. Patients also receive zoledronic acid IV over 15-30 minutes at 28 days prior to stem cell transplantation and at 3 and 6 months after transplantation.
Period: Overall Study
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Started | 29 | 32
Completed | 19 | 11
Not Completed | 10 | 21
Not completed — Death | 3 | 6
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Early relapse | 2 | 8
Not completed — Missing data | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa) | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 32 | 61
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10) | 51 (12) | 51 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 16 | 23 | 39
Region of Enrollment [Number; unit: participants]
  United States | 29 | 32 | 61

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Bone Mineral Density
Description: Change in bone mineral density of the femoral neck measured from baseline to 12 months after transplant utilizing Dual-energy X-ray absorptiometry (DEXA) scan. Comparison of difference between the standard of care group (receiving calcium and vitamin D)and the Zometa group. The measurement consists of baseline bone mineral density measurements with followup measurements at 12 months.
  This will be analyzed as a continuous variable. Percent change in bone mineral density (BMD) will be calculated as (BMD change) x 100/BMD baseline.
Time Frame: From Time of Transplant to 12 Months Post-Transplant
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Arm II (Treatment With Zometa): Patients receive vitamin D and calcium as in arm I. Patients also receive zoledronic acid intravenously (IV) over 15-30 minutes at 28 days prior to stem cell transplantation and at 3 and 6 months after transplantation.
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Number analyzed (Participants) | 29 | 32
percent | -0.0714 (0.101) | -0.0036 (0.089)

2. Secondary Outcome: Mean Change in Serum Osteocalcin
Description: Change in bone resorption markers of bone metabolism measured at baseline and 12 months post transplant for all enrolled patients. As osteocalcin is produced by osteoblasts, it is often used as a marker for the bone formation process.
Time Frame: From Time of Transplant to 12 Months Post-Transplant
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Arm II (Treatment With Zometa): Patients receive vitamin D and calcium as in arm I. Patients also receive zoledronic acid intravenously (IV)( over 15-30 minutes at 28 days prior to stem cell transplantation and at 3 and 6 months after transplantation.
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Number analyzed (Participants) | 29 | 32
ng/ml | -3.6 (24.1) | -11.3 (7.6)

3. Secondary Outcome: Mean Change in Serum Bone Specific Alkaline Phosphate
Description: Change in bone resorption markers of bone metabolism measured at baseline and 12 months post transplant for all enrolled patients. The decrease in serum bone-specific alkaline phosphatase predicts bone mineral density response to hormone replacement therapy in early postmenopausal women.
Time Frame: From Time of Transplant to 12 Months Post-Transplant
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Number analyzed (Participants) | 29 | 32
U/L | -3.0 (5.7) | -4.3 (5.6)

4. Secondary Outcome: Mean Change in Urinary N-terminal Telopeptide
Description: Change in bone resorption markers of bone metabolism measured at baseline and 12 months post transplant for all enrolled patients. In bone physiology, the N-terminal telopeptide is a biomarker used to measure the rate of bone turnover.
Time Frame: From Time of Transplant to 12 Months Post-Transplant
Measure: Mean (Standard Deviation); unit: nM Bone Collagen Equivalents/mM creatini
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Number analyzed (Participants) | 29 | 32
nM Bone Collagen Equivalents/mM creatini | -22.5 (137.7) | -103.0 (137.7)

5. Secondary Outcome: Mean Change in Luteinizing Hormone
Description: Change in bone resorption markers of bone metabolism measured at baseline and 12 months post transplant for all enrolled patients. Luteinizing hormone is a hormone produced by the anterior pituitary gland.
Time Frame: From Time of Transplant to 12 Months Post-Transplant
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Number analyzed (Participants) | 29 | 32
IU/L | 18.8 (21.6) | 12.8 (16.8)

6. Secondary Outcome: Mean Change in Follicle-Stimulating Hormone
Description: Change in bone resorption markers of bone metabolism measured at baseline and 12 months post transplant for all enrolled patients. Follicle-stimulating hormone is a hormone produced by the anterior pituitary gland.
Time Frame: From Time of Transplant to 12 Months Post-Transplant
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Number analyzed (Participants) | 29 | 32
IU/L | 14.0 (46.7) | 6.6 (6.5)

7. Secondary Outcome: Mean Change in Thyroid Function Test 4
Description: Change in bone resorption markers of bone metabolism measured at baseline and 12 months post transplant for all enrolled patients. Individuals who have hyperthyroidism will have an elevated thyroxine (FT4). Low serum thyroxine can also indicate a pituitary problem.
Time Frame: From Time of Transplant to 12 Months Post-Transplant
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Number analyzed (Participants) | 29 | 32
ng/dL | -0.6 (2.2) | -0.2 (0.9)

8. Secondary Outcome: Mean Change in Ultrasensitive Estradiol
Description: Change in bone resorption markers of bone metabolism measured at baseline and 12 months post transplant for all enrolled patients. In women estradiol is responsible for growth of the breast and reproductive epithelia, maturation of long bones and development of the secondary sexual characteristics.
Time Frame: From Time of Transplant to 12 Months Post-Transplant
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Number analyzed (Participants) | 29 | 32
pg/ml | -3.6 (19.4) | -6.3 (21.0)

9. Secondary Outcome: Mean Change in Total Testosterone
Description: Change in bone resorption markers of bone metabolism measured at baseline and 12 months post transplant for all enrolled patients. Testosterone affects the brain, bone and muscle mass, fat distribution, the vascular system, energy levels, genital tissues, and sexual functioning.
Time Frame: From Time of Transplant to 12 Months Post-Transplant
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Number analyzed (Participants) | 29 | 32
ng/dL | -65.4 (130.4) | -23.6 (140.0)

ADVERSE EVENTS:
Time Frame: Serious adverse events are collected from first dose of study medication through 30 days of the last dose of treatment. Any death that occured within one year of first treatment is also included.
Description: Adverse reactions to Zometa® (zoledronic acid for injection) are usually mild and transient and similar to those reported for other bisphosphonates. Therefore, only serious events were collected.
Arm/Group | Arm I (Standard of Care) | Arm II (Treatment With Zometa)
Serious Adverse Events (participants affected / at risk) | 8/29 | 21/32
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Standard of Care) (N=29) | Arm II (Treatment With Zometa) (N=32)
Death (General disorders) | 6 (6) | 15 (15)
Graft-versus-host disease (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Idiopathic pulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection with unknown absolute neutrophil count (Infections and infestations) | 0 (0) | 2 (2) — Pneumonia
New Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nosebleed (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pseudomonas sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes